CLINICAL TRIAL: NCT01771146
Title: A Prospective Evaluation of Neoadjuvant FOLFIRINOX Regimen in Patients With Non-metastatic Pancreas Cancer (Baylor University Medical Center and Texas Oncology Experience)
Brief Title: Neoadjuvant FOLFIRINOX Regimen in Patients With Non-metastatic Pancrease Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012-180
Record Dates: First submitted 2013-01-08; First posted 2013-01-18 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pancreas Cancer; Localized Pancreas Cancer; Non-metastatic Pancreas Cancer
Keywords: Non-metastatic Pancreas Cancer; Pancreatic Cancer; Cancer of Pancreas; Adenocarcinoma of Pancreas; Neoadjuvant
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant FOLFIRINOX Regimen (Other): Single arm, treated with neoadjuvant FOLFIRINOX prior to surgical resection
  Interventions: Drug: FOLFIRINOX Regimen

INTERVENTIONS:
Drug: FOLFIRINOX Regimen — 6 cycles of FOLFIRINOX prior to surgical resection: Eloxatin® (Oxaliplatin) 85 mg per square meter 2-hour IV infusion Camptosar® (Irinotecan Hydrochloride) 180 mg per square meter 90-minute IV infusion via Y-connector adrucil (Fluorouracil; 5-FU)2400 mg per square meter 46-hour IV infusion
  Other Names: FOLFIRINOX; Oxaliplatin; Irinotecan; 5-FU; Eloxatin; Camptosar; Adrucil

SUMMARY:
A prospective evaluation of neoadjuvant FOLFIRINOX regimen in patients with non-metastatic pancreas cancer (Baylor University Medical Center and Texas Oncology Experience)

DETAILED DESCRIPTION:
Patients with pancreas cancer will be enrolled and treated with a planned course of 6 cycles (3 months) of chemotherapy with FOLFIRINOX prior to undergoing surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or non-pregnant and non-lactating female
* Histologically or cytologically confirmed adenocarcinoma of pancreas
* Patients must have satisfactory blood counts and blood chemistry levels at baseline (refer to Appendix 2, Study Laboratory References Range).
* Patient has Eastern Cooperative Oncology Group(ECOG) Performance Status 0 to 1 (refer to Appendix 7):
* 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
* 1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
* Signed study consent form

Exclusion Criteria:

* <18 years of age
* Pregnant or lactating female
* Patient has islet cell neoplasms
* Patient has known brain metastases
* Patient has metastatic disease
* Active secondary malignancies
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known infection with hepatitis B, hepatitis C, or cirrhosis
* Major surgery or vascular device placement (excluding ports for IV medication/chemotherapy) within 2 weeks prior to Day 1 of treatment in study
* Prior chemotherapy or radiation for pancreatic cancer
* History of allergy or hypersensitivity to the study drugs
* Patient is enrolled in any outside (outside Baylor University Medical Center or Texas Oncology) clinical protocol or investigational trial
* Significant cardiac disease as defined as New York Heart Association (NYHA) classification III or IV, uncontrolled congestive heart failure (CHF), or prior myocardial infarction (MI) last 6-months
* Any prior gastrointestinal (GI) disease or history of prior pelvic or abdominal radiation which in the opinion of the investigator may place the patient at increased risk
* Peripheral sensory neuropathy ≥ to grade 2 at baseline
* Significant co-morbidities deemed by investigator as unsuitable for participation/enrollment
* Study consent form not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as defined by the length of time that a patient survives without any signs or symptoms of that cancer or any other type of cancer | Up to 5 years

SECONDARY OUTCOMES:
• The length of time from diagnosis (enrollment) to death | Up to 5 years
• Overall Survival rate defined by the % of people who are alive for a certain period of time after diagnosis | Up to 5 years
• R0 resection as defined as microscopically negative margins | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Celinski, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center - Texas Oncology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided